CLINICAL TRIAL: NCT00593047
Title: A Phase II, Placebo-Controlled, Double-Blind, Randomised, 12-Week, Parallel-Group Study to Assess the Efficacy of Different Doses of KB2115 as Add on to Statin Treatment in Patients With Dyslipidemia
Brief Title: LDL-Cholesterol Lowering Effect of KB2115 as Add on to Statin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karo Bio AB (Industry)
Responsible Party: Dr Jens Kristensen, Chief Medical Officer, Karo Bio AB
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBT004; 2007-004413-33
Record Dates: First submitted 2007-12-17; First posted 2008-01-14 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-05

CONDITIONS: Dyslipidemia
Keywords: hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — 3-((3,5-dibromo-4-(4-hydroxy-3-(1-methylethyl)phenoxy)phenyl)amino)-3-oxopropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Statin + placebo
  Interventions: Drug: KB2115
- 2 (Experimental): Statin + KB2115 dose 1
  Interventions: Drug: KB2115
- 3 (Experimental): Statin + KB2115 dose 2
  Interventions: Drug: KB2115
- 4 (Experimental): Statin + KB2115 dose 3
  Interventions: Drug: KB2115

INTERVENTIONS:
Drug: KB2115 — tablet formulation given once daily for 12 weeks

SUMMARY:
Thyroid hormones are known to reduce cholesterol levels through regulation of a number of key enzymes involved in synthesis, degradation, and lipid transport. However, the currently marketed thyroid agonists are non-selective, and cannot be used for the treatment of hypercholesterolemia due to extrahepatic consequences of hyperthyroidism, especially on heart, bone, and muscle.

To take advantage of thyroid hormone effect on lipid metabolism for the treatment of hypercholesterolemia, it is necessary to develop a selective thyroid receptor agonist that can induce hyperthyroidism in the liver, while an euthyroid state is preserved in the extrahepatic tissue. KB2115 is a thyroid agonist developed to be liver selective.

The purpose of the study is to assess the efficacy and safety of KB2115 as add on therapy to low and middle doses of statin following 12 weeks of exposure compared to placebo. The aim of the study is to assess efficacy (LDL-cholesterol lowering effects) and safety of KB2115 at doses between 25 and 100 µg and to define a clinically relevant dose or dose range for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Males or females aged 18 to 75 years. Female patients must be non-fertile. To be considered as non-fertile, females must fulfil the following:

   * Non-nursing and non-pregnant 12 months prior to enrolment
   * Not of child bearing potential ie, either documented irreversible surgically sterile (bilateral oophorectomy or hysterectomy is acceptable, but not tubal ligation) or post-menopausal. Post-menopausal is defined as serum follicle-stimulating hormone (FSH) levels in the post-menopausal range combined with amenorrhea for more than 1 year in a woman above 50 years of age, or amenorrhea for more than 2 years below 50 years of age
3. Patients with hypercholesterolemia treated with stable doses of the below listed lipid lowering medication for at least 3 months prior to randomization

   * Atorvastatin not more than 20 mg/day or
   * Simvastatin not more than 40 mg/day
4. LDL-cholesterol > 3.0 mmol/L (Week -1)
5. Subject able and willing to comply with all study requirements
6. At randomization, diet as instructed by the investigator during the last 4 weeks prior to randomization and willingness to follow these instructions throughout the study

Exclusion Criteria:

1. Cholesterol lowering agents other than the defined statins
2. History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study as judged by the investigator
3. Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product as judged by the investigator
4. Chronic (> 3 months) pain condition requiring daily medication with pain killers
5. Glycosylated haemoglobin (HbA1c) > 7.0%
6. Diabetes requiring medication other than metformin
7. Clinically abnormal physical findings and laboratory values as judged by the investigator and abnormal resting ECG, eg, QTc interval > 450 msec
8. Body Mass Index of ≥ 40 kg/m2
9. Resent history (< 3 month) of stroke or transient ischemic attacks
10. History of seizure disorder, except febrile convulsions
11. A current diagnosis of cancer, unless in remission
12. Blood pressure (BP) of > 160/95 mm Hg
13. History of cardiac arrhythmia, such as intermittent supraventricular tachyarrhythmia and atrial fibrillation
14. Unstable angina pectoris, myocardial infarction or coronary bypass graft surgery or percutaneous coronary intervention < 6 month before randomization
15. Congestive heart failure New York Heart Association Class > 2
16. Unstable or severe angina pectoris or peripheral artery disease
17. Known thyroid disease or thyroid biomarkers (TSH, T3, free T3, T4, free T4) outside reference range for normal at enrolment and at baseline
18. Positive urine pregnancy test in women at enrolment
19. Use of thyroid replacement therapy and hormone replacement therapy (including contraceptive pills) for last 3 months before randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 12 weeks

SECONDARY OUTCOMES:
Triglyceride | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kristensen, MD, PhD, Study Director — Karo Bio AB
Locations (1):
- Carl-Peter Anderberg, Gothemburg, Sweden

REFERENCES:
- [Derived] Ladenson PW, Kristensen JD, Ridgway EC, Olsson AG, Carlsson B, Klein I, Baxter JD, Angelin B. Use of the thyroid hormone analogue eprotirome in statin-treated dyslipidemia. N Engl J Med. 2010 Mar 11;362(10):906-16. doi: 10.1056/NEJMoa0905633. PMID 20220185